CLINICAL TRIAL: NCT00652951
Title: Non-inferiority of Co-administration of GSK Biologicals'Pneumococcal Conjugate Vaccine GSK1024850A With DTPa-IPV-Hib Versus Co-administration With DTPa-HBV-IPV/Hib.
Brief Title: Co-administration of Pneumococcal Conjugate Vaccine With DTPa-IPV-Hib Versus Co-administration With DTPa-HBV-IPV/Hib
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 110142; 111053; 2007-004002-26 (EudraCT Number)
Record Dates: First submitted 2008-03-21; First posted 2008-04-04 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Infections, Streptococcal
MeSH Terms: conditions — Streptococcal Infections | interventions — PHiD-CV vaccine; diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Synflorix + Infanrix hexa Group (Active Comparator): Subjects received 3 doses of SynflorixTM vaccine co-administered with Infanrix hexaTM at 2, 3 and 4 months of age (Study Months 0, 1, 2) and received a booster dose of each vaccine between 11 and 13 months of age (Study Month 9). All vaccines were administered intramuscularly in the right (SynflorixTM) or left (Infanrix hexaTM) thigh or deltoid.
  Interventions: Biological: GSK Biologicals´ Pneumococcal Conjugate Vaccine GSK1024850A (Synflorix™); Biological: Infanrix™ hexa.
- Synflorix + Pediacel Group (Experimental): Subjects received 3 doses of SynflorixTM vaccine co-administered with PediacelTM at 2, 3 and 4 months of age (Study Months 0, 1, 2) and received a booster dose of each vaccine between 11 and 13 months of age (Study Month 9). All vaccines were administered intramuscularly in the right (SynflorixTM) or left (PediacelTM) thigh or deltoid.thigh or deltoid.
  Interventions: Biological: GSK Biologicals´ Pneumococcal Conjugate Vaccine GSK1024850A (Synflorix™); Biological: Pediacel™
- Prevenar + Pediacel Group (Active Comparator): Subjects received 3 doses of PrevenarTM co-administered with PediacelTM vaccine at 2, 3 and 4 months of age (Study Months 0, 1, 2) and received a booster dose of each vaccine between 11 and 13 months of age (Study Month 9). All vaccines were administered intramuscularly in the right (PrevenarTM) or left (PediacelTM) thigh or deltoid.
  Interventions: Biological: Pediacel™; Biological: Prevenar™

INTERVENTIONS:
Biological: GSK Biologicals´ Pneumococcal Conjugate Vaccine GSK1024850A (Synflorix™) — Intramuscular injection, 3 doses in the primary vaccination and 1 dose in the booster vaccination
  Arms: Synflorix + Infanrix hexa Group; Synflorix + Pediacel Group
Biological: Infanrix™ hexa. — Intramuscular injection, , 3 doses in the primary vaccination and 1 dose in the booster vaccination
  Arms: Synflorix + Infanrix hexa Group
Biological: Pediacel™ — Intramuscular injection, , 3 doses in the primary vaccination and 1 dose in the booster vaccination
  Arms: Prevenar + Pediacel Group; Synflorix + Pediacel Group
Biological: Prevenar™ — Intramuscular injection, , 3 doses in the primary vaccination and 1 dose in the booster vaccination
  Arms: Prevenar + Pediacel Group

SUMMARY:
The purpose of this trial is to evaluate the immunogenicity and safety of a pneumococcal conjugate vaccine when co-administered with DTPa-IPV-Hib or DTPa-HBV-IPV/Hib in infants as a three-dose primary immunisation course during the first 6 months of life and as a booster dose at 11-12 months of age. The impact of the pneumococcal conjugate vaccine on nasopharyngeal carriage of S. pneumoniae and H. influenzae in children in their first two years of life will also be assessed. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardian(s) can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits) should be enrolled in the study.
* A male or female between, and including, 6-12 weeks (42-90 days) of age at the time of the first vaccination.
* Written informed consent obtained from both parents or from the guardian(s) of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of at least 36 weeks.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the entire study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting from one month (30 days) before and up to one month (30 days) after each dose of study vaccine.
* Previous vaccination against diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b and/or Streptococcus pneumoniae.
* Children for whom hepatitis B vaccination is required according to the local recommendations
* History of or intercurrent diphtheria, tetanus, pertussis, hepatitis B, polio, Haemophilus influenzae type b disease.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 780 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2009-05-12 (Actual); Study Completion 2010-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hoofddorp, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] van den Bergh MR, Spijkerman J, Francois N, Swinnen K, Borys D, Schuerman L, Veenhoven RH, Sanders EA. Immunogenicity, safety, and reactogenicity of the 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine and DTPa-IPV-Hib when coadministered as a 3-dose primary vaccination schedule in The Netherlands: a randomized controlled trial. Pediatr Infect Dis J. 2011 Sep;30(9):e170-8. doi: 10.1097/INF.0b013e31821a0614. PMID 21487327
- [Background] van den Bergh MR, Spijkerman J, Swinnen KM, Francois NA, Pascal TG, Borys D, Schuerman L, Ijzerman EP, Bruin JP, van der Ende A, Veenhoven RH, Sanders EA. Effects of the 10-valent pneumococcal nontypeable Haemophilus influenzae protein D-conjugate vaccine on nasopharyngeal bacterial colonization in young children: a randomized controlled trial. Clin Infect Dis. 2013 Feb;56(3):e30-9. doi: 10.1093/cid/cis922. Epub 2012 Nov 1. PMID 23118268
- [Background] van den Bergh MR, Spijkerman J, Francois N, Swinnen K, Borys D, Schuerman L, Veenhoven RH, Sanders EA. Immunogenicity, Safety and Reactogenicity of a Booster Dose of the 10-Valent Pneumococcal Nontypeable H. influenzae Protein D Conjugate Vaccine Coadministered With DTPa-IPV-Hib in Dutch Children: A Randomized Controlled Trial. Pediatr Infect Dis J. 2016 Jul;35(7):e206-19. doi: 10.1097/INF.0000000000001170. PMID 27097348
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 110142 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 110142 are summarised with study 111053 on GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110142 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110142 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110142 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110142 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110142 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110142 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included a Primary (PRI) Phase, up to Month 3, followed by a Booster (BST) Phase, up to Month 9.
Pre-assignment Details: At screening the following was performed: informed consent was obtained and signed from subjects' parents/guardians, check for inclusion/exclusion criteria and contraindications/precautions was performed as regards to vaccination, and medical history of subjects was collected. Subjects' pre-vaccination body temperature was evaluated.
Groups:
- Synflorix + Infanrix Hexa Group: Subjects received 3 doses of Synflorix vaccine co-administered with Infanrix hexa at 2, 3 and 4 months of age (Study Months 0, 1, 2) and received a booster dose of each vaccine between 11 and 13 months of age (Study Month 9). All vaccines were administered intramuscularly in the right (Synflorix) or left (Infanrix hexa) thigh or deltoid.
- Synflorix + Pediacel Group: Subjects received 3 doses of Synflorix vaccine co-administered with Pediacel at 2, 3 and 4 months of age (Study Months 0, 1, 2) and received a booster dose of each vaccine between 11 and 13 months of age (Study Month 9). All vaccines were administered intramuscularly in the right (Synflorix) or left (Pediacel) thigh or deltoid.
- Prevenar + Pediacel Group: Subjects received 3 doses of Prevenar co-administered with Pediacel vaccine at 2, 3 and 4 months of age (Study Months 0, 1, 2) and received a booster dose of each vaccine between 11 and 13 months of age (Study Month 9). All vaccines were administered intramuscularly in the right (Prevenar) or left (Pediacel) thigh or deltoid.
Period: Primary Phase
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Started | 260 | 260 | 260
Completed | 260 | 260 | 260
Not Completed | 0 | 0 | 0
Period: Booster Phase
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Started | 257 | 259 | 258
Completed | 256 | 258 | 258
Not Completed | 1 | 1 | 0
Not completed — Adverse event, non-fatal | 0 | 1 | 0
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group | Total
Number analyzed (Participants) | 260 | 260 | 260 | 780
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 7.4 (1.2) | 7.6 (1.29) | 7.6 (1.26) | 7.53 (1.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 130 | 136 | 384
  Male | 142 | 130 | 124 | 396
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African heritage/African American | 0 | 1 | 0 | 1
  Geographic ancestry: Asian - Central/South Asian heritage | 0 | 0 | 1 | 1
  Geographic ancestry: White - Arabic/North African heritage | 0 | 1 | 0 | 1
  Geographic ancestry: White - Caucasian/European heritage | 258 | 255 | 256 | 769
  Geographic ancestry: Unspecified | 2 | 3 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Antibody Concentrations Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Anti-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F) - Primary Vaccination
Description: Anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations (Anti-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F) were measured by 22F-inhibition Enzyme-Linked ImmunSorbent Assay (ELISA); presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (μg/mL). The seropositivity cut-off for the assay was greater than or equal to (≥) 0.05 μg/mL.
Time Frame: At Month 3, one month after the administration of the third dose of pneumococcal conjugate vaccine
Population: The Primary ATP cohort for immunogenicity included all evaluable subjects for whom data concerning immunogenicity outcome measures were available. This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component post-dose III.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 194 | 189 | 192
μg/mL
  Anti-1: number analyzed (Participants) | 181 | 178 | 178
  Anti-1 | 1.17 [1.02 to 1.33] | 1.31 [1.16 to 1.48] | 0.03 [0.03 to 0.03]
  Anti-4: number analyzed (Participants) | 192 | 185 | 191
  Anti-4 | 1.61 [1.41 to 1.84] | 1.59 [1.38 to 1.83] | 2.44 [2.19 to 2.73]
  Anti-5: number analyzed (Participants) | 187 | 181 | 178
  Anti-5 | 2.11 [1.88 to 2.37] | 2.16 [1.92 to 2.43] | 0.03 [0.03 to 0.03]
  Anti-6B: number analyzed (Participants) | 177 | 174 | 180
  Anti-6B | 0.33 [0.26 to 0.4] | 0.35 [0.28 to 0.43] | 0.41 [0.34 to 0.51]
  Anti-7F: number analyzed (Participants) | 192 | 187 | 183
  Anti-7F | 1.7 [1.52 to 1.9] | 1.77 [1.57 to 1.99] | 0.04 [0.03 to 0.04]
  Anti-9V: number analyzed (Participants) | 185 | 186 | 187
  Anti-9V | 1.4 [1.2 to 1.63] | 1.47 [1.29 to 1.68] | 2.14 [1.91 to 2.4]
  Anti-14: number analyzed (Participants) | 192 | 187 | 192
  Anti-14 | 3.38 [2.99 to 3.81] | 3.33 [2.93 to 3.78] | 3.64 [3.24 to 4.1]
  Anti-18C: number analyzed (Participants) | 194 | 189 | 191
  Anti-18C | 1.73 [1.45 to 2.05] | 1.07 [0.92 to 1.25] | 2.1 [1.83 to 2.4]
  Anti-19F: number analyzed (Participants) | 189 | 183 | 189
  Anti-19F | 2.07 [1.73 to 2.48] | 1.96 [1.64 to 2.34] | 3.04 [2.71 to 3.42]
  Anti-23F: number analyzed (Participants) | 179 | 175 | 184
  Anti-23F | 0.5 [0.41 to 0.6] | 0.54 [0.44 to 0.66] | 1.24 [1.04 to 1.47]
Statistical Analysis 1: Comparison: Synflorix + Infanrix Hexa Group vs Synflorix + Pediacel Group; The 2-sided 95% confidence interval (CI) of the geometric mean concentration (GMC) ratio between the Synflorix + Infanrix hexa and Synflorix + Pediacel groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), at one month after Dose 3 of pneumococcal vaccine, was computed for each of the 10 pneumococcal vaccine serotypes and protein D. This statistical method concerns pneumococcal vaccine serotype 1; Test type: Non-Inferiority — Non-inferiority criteria: The upper limit (UL) of the 2-sided 95% confidence interval (CI) of the GMC ratio for between groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), was lower than 2 for the pneumococcal vaccine serotype 1; ANOVA; GMC ratio = 0.89, 95% CI 2-sided [0.74 to 1.07]
Statistical Analysis 2: Comparison: Synflorix + Infanrix Hexa Group vs Synflorix + Pediacel Group; The 2-sided 95% CI of the geometric mean concentration (GMC) ratio between the Synflorix + Infanrix hexa and Synflorix + Pediacel groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), at one month after Dose 3 of pneumococcal vaccine, was computed for each of the 10 pneumococcal vaccine serotypes and protein D. This statistical method concerns pneumococcal vaccine serotype 4; Test type: Non-Inferiority — Non-inferiority criteria: The upper limit (UL) of the 2-sided 95% CI of the GMC ratio for between groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), was lower than 2 for the pneumococcal vaccine serotype 4; ANOVA; GMC ratio = 1.01, 95% CI 2-sided [0.84 to 1.23]
Statistical Analysis 3: Comparison: Synflorix + Infanrix Hexa Group vs Synflorix + Pediacel Group; The 2-sided 95% CI of the geometric mean concentration (GMC) ratio between the Synflorix + Infanrix hexa and Synflorix + Pediacel groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), at one month after Dose 3 of pneumococcal vaccine, was computed for each of the 10 pneumococcal vaccine serotypes and protein D. This statistical method concerns pneumococcal vaccine serotype 5; Test type: Non-Inferiority — Non-inferiority criteria: The upper limit (UL) of the 2-sided 95% CI of the GMC ratio for between groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), was lower than 2 for the pneumococcal vaccine serotype 5; ANOVA; GMC ratio = 0.98, 95% CI 2-sided [0.83 to 1.15]
Statistical Analysis 4: Comparison: Synflorix + Infanrix Hexa Group vs Synflorix + Pediacel Group; The 2-sided 95% CI of the geometric mean concentration (GMC) ratio between the Synflorix + Infanrix hexa and Synflorix + Pediacel groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), at one month after Dose 3 of pneumococcal vaccine, was computed for each of the 10 pneumococcal vaccine serotypes and protein D. This statistical method concerns pneumococcal vaccine serotype 6B; Test type: Non-Inferiority — Non-inferiority criteria: The upper limit (UL) of the 2-sided 95% CI of the GMC ratio for between groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), was lower than 2 for the pneumococcal vaccine serotype 6B; ANOVA; GMC ratio = 0.93, 95% CI 2-sided [0.69 to 1.26]
Statistical Analysis 5: Comparison: Synflorix + Infanrix Hexa Group vs Synflorix + Pediacel Group; The 2-sided 95% CI of the geometric mean concentration (GMC) ratio between the Synflorix + Infanrix hexa and Synflorix + Pediacel Group groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), at one month after Dose 3 of pneumococcal vaccine, was computed for each of the 10 pneumococcal vaccine serotypes and protein D. This statistical method concerns pneumococcal vaccine serotype 7F; Test type: Non-Inferiority — Non-inferiority criteria: The upper limit of the 2-sided 95% CI of the GMC ratio for between groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group Group), was lower than 2 for the pneumococcal vaccine serotype 7F; ANOVA; GMC ratio = 0.96, 95% CI 2-sided [0.82 to 1.13]
Statistical Analysis 6: Comparison: Synflorix + Infanrix Hexa Group vs Synflorix + Pediacel Group; The 2-sided 95% CI of the geometric mean concentration (GMC) ratio between the Synflorix + Infanrix hexa and Synflorix + Pediacel groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), at one month after Dose 3 of pneumococcal vaccine, was computed for each of the 10 pneumococcal vaccine serotypes and protein D. This statistical method concerns pneumococcal vaccine serotype 9V; Test type: Non-Inferiority — Non-inferiority criteria: The upper limit (UL) of the 2-sided 95% CI of the GMC ratio for between groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), was lower than 2 for the pneumococcal vaccine serotype 9V; ANOVA; GMC ratio = 0.95, 95% CI 2-sided [0.78 to 1.16]
Statistical Analysis 7: Comparison: Synflorix + Infanrix Hexa Group vs Synflorix + Pediacel Group; The 2-sided 95% CI of the geometric mean concentration (GMC) ratio between the Synflorix + Infanrix hexa and Synflorix + Pediacel groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), at one month after Dose 3 of pneumococcal vaccine, was computed for each of the 10 pneumococcal vaccine serotypes and protein D. This statistical method concerns pneumococcal vaccine serotype 14; Test type: Non-Inferiority — Non-inferiority criteria: The upper limit (UL) of the 2-sided 95% CI of the GMC ratio for between groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), was lower than 2 for the pneumococcal vaccine serotype 14; ANOVA; GMC ratio = 1.01, 95% CI 2-sided [0.85 to 1.21]
Statistical Analysis 8: Comparison: Synflorix + Infanrix Hexa Group vs Synflorix + Pediacel Group; The 2-sided 95% CI of the geometric mean concentration (GMC) ratio between the Synflorix + Infanrix hexa and Synflorix + Pediacel groups (Synflorix + Infanrix hexa Group over ), at one month after Dose 3 of pneumococcal vaccine, was computed for each of the 10 pneumococcal vaccine serotypes and protein D. This statistical method concerns pneumococcal vaccine serotype 18C; Test type: Non-Inferiority — Non-inferiority criteria: The upper limit (UL) of the 2-sided 95% CI of the GMC ratio for between groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), was lower than 2 for the pneumococcal vaccine serotype 18C; ANOVA; GMC ratio = 1.61, 95% CI 2-sided [1.28 to 2.03]
Statistical Analysis 9: Comparison: Synflorix + Infanrix Hexa Group vs Synflorix + Pediacel Group; The 2-sided 95% CI of the geometric mean concentration (GMC) ratio between the Synflorix + Infanrix hexa and Synflorix + Pediacel groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), at one month after Dose 3 of pneumococcal vaccine, was computed for each of the 10 pneumococcal vaccine serotypes and protein D. This statistical method concerns pneumococcal vaccine serotype 19F; Test type: Non-Inferiority — Non-inferiority criteria: The upper limit (UL) of the 2-sided 95% CI of the GMC ratio for between groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), was lower than 2 for the pneumococcal vaccine serotype 19F; ANOVA; GMC ratio = 1.06, 95% CI 2-sided [0.82 to 1.36]
Statistical Analysis 10: Comparison: Synflorix + Infanrix Hexa Group vs Synflorix + Pediacel Group; The 2-sided 95% CI of the geometric mean concentration (GMC) ratio between the Synflorix + Infanrix hexa Group and Synflorix + Pediacel groups (Synflorix + Infanrix hexa Group Group over Synflorix + Pediacel Group), at one month after Dose 3 of pneumococcal vaccine, was computed for each of the 10 pneumococcal vaccine serotypes and protein D. This statistical method concerns pneumococcal vaccine serotype 23F; Test type: Non-Inferiority — Non-inferiority criteria: The upper limit (UL) of the 2-sided 95% CI of the GMC ratio for between groups (Synflorix + Infanrix hexa Group Group over Synflorix + Pediacel Group), was lower than 2 for the pneumococcal vaccine serotype 23F; ANOVA; GMC ratio = 0.92, 95% CI 2-sided [0.7 to 1.23]

2. Primary Outcome: Antibody Concentration Against Protein D (PD) - Primary Vaccination
Description: Anti-PD antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in ELISA units per milliliter (EL.U/mL). The seropositivity cut-off for the assay was ≥ 100 EL.U/mL.
Time Frame: At Month 3, one month after the administration of the third dose of pneumococcal conjugate vaccine
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 195 | 189 | 182
EL.U/mL | 1580 [1409.5 to 1771.1] | 1743 [1560.2 to 1947.2] | 69.7 [63 to 77.1]
Statistical Analysis 1: Comparison: Synflorix + Infanrix Hexa Group vs Synflorix + Pediacel Group; The 2-sided 95% CI of the geometric mean concentration (GMC) ratio between the Synflorix + Infanrix hexa and Synflorix + Pediacel groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), at one month after Dose 3 of pneumococcal vaccine, was computed for each of the 10 pneumococcal vaccine serotypes and protein D. This statistical method concerns protein D; Test type: Non-Inferiority — Non-inferiority criteria: The upper limit (UL) of the 2-sided 95% CI of the GMC ratio for between groups (Synflorix + Infanrix hexa Group over Synflorix + Pediacel Group), was lower than 2 for protein D; ANOVA; GMC ratio = 0.91, 95% CI 2-sided [0.77 to 1.06]

3. Secondary Outcome: Number of Subjects With Antibody Concentrations Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Anti-1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) ≥ 0.2 μg/mL - Primary Vaccination
Description: Antibody concentrations against the pneumococcal serotypes were assessed by 22F-inhibition ELISA. The reference cut-off value of the assay was an antibody concentration greater than or equal to (≥) 0.02 µg/mL.
Time Frame: At Month 3, one month after the administration of the third vaccine dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 194 | 189 | 192
Participants
  Anti-1: number analyzed (Participants) | 181 | 178 | 178
  Anti-1 | 174 | 176 | 5
  Anti-4: number analyzed (Participants) | 192 | 185 | 191
  Anti-4 | 188 | 180 | 189
  Anti-5: number analyzed (Participants) | 187 | 181 | 178
  Anti-5 | 187 | 179 | 0
  Anti-6B: number analyzed (Participants) | 177 | 174 | 180
  Anti-6B | 122 | 113 | 124
  Anti-7F: number analyzed (Participants) | 192 | 187 | 183
  Anti-7F | 190 | 186 | 11
  Anti-9V: number analyzed (Participants) | 185 | 186 | 187
  Anti-9V | 176 | 181 | 184
  Anti-14: number analyzed (Participants) | 192 | 187 | 192
  Anti-14 | 191 | 187 | 192
  Anti-18C: number analyzed (Participants) | 194 | 189 | 191
  Anti-18C | 183 | 178 | 187
  Anti-19F: number analyzed (Participants) | 189 | 183 | 189
  Anti-19F | 180 | 174 | 189
  Anti-23F: number analyzed (Participants) | 179 | 175 | 184
  Anti-23F | 134 | 133 | 171

4. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F - Primary Vaccination
Description: Titers were presented as geometric mean titers (GMTs), for the seropositivity cut-off value of 8.
Time Frame: At Month 3, one month after the administration of the third vaccine dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 139 | 135 | 132
Titers
  Opsono-1: number analyzed (Participants) | 132 | 126 | 125
  Opsono-1 | 20.7 [15.6 to 27.6] | 20.8 [15.8 to 27.4] | 4.7 [4.1 to 5.2]
  Opsono-4: number analyzed (Participants) | 133 | 132 | 129
  Opsono-4 | 592.9 [475.9 to 738.7] | 600.4 [492.2 to 732.3] | 838.4 [718.7 to 978.2]
  Opsono-5: number analyzed (Participants) | 138 | 134 | 132
  Opsono-5 | 54.8 [44 to 68.4] | 60.1 [48.2 to 74.8] | 4.2 [3.9 to 4.6]
  Opsono-6B: number analyzed (Participants) | 129 | 130 | 123
  Opsono-6B | 261.3 [176 to 388] | 296.4 [198 to 443.7] | 633 [419 to 956.4]
  Opsono-7F: number analyzed (Participants) | 130 | 127 | 114
  Opsono-7F | 2063.3 [1691.7 to 2516.6] | 2136.1 [1707.9 to 2671.5] | 18.4 [12.1 to 28]
  Opsono-9V: number analyzed (Participants) | 132 | 129 | 125
  Opsono-9V | 863.6 [687.6 to 1084.7] | 1277.7 [1053.3 to 1550.1] | 1194 [1009.5 to 1412.1]
  Opsono-14: number analyzed (Participants) | 134 | 135 | 127
  Opsono-14 | 990.4 [820.6 to 1195.5] | 1086.4 [899.6 to 1311.9] | 1373.3 [1040.4 to 1812.7]
  Opsono-18C: number analyzed (Participants) | 133 | 129 | 129
  Opsono-18C | 122.6 [89.4 to 168.2] | 84.2 [60.9 to 116.5] | 213.6 [163.6 to 278.8]
  Opsono-19F: number analyzed (Participants) | 137 | 133 | 130
  Opsono-19F | 133 [98.1 to 180.2] | 143.8 [108.6 to 190.3] | 39.2 [30.6 to 50.4]
  Opsono-23F: number analyzed (Participants) | 139 | 133 | 130
  Opsono-23F | 847.4 [626.5 to 1146.3] | 1089 [800.2 to 1482] | 3703.4 [3119.4 to 4396.8]

5. Secondary Outcome: Number of Subjects With Antibody Concentrations Against Pneumococcal Cross-reactive Serotypes 6A and 19A (Anti-6A and 19A) ≥ 0.2 μg/mL - Primary Vaccination.
Description: Antibody concentrations against the cross- reactive pneumococcal serotypes were assessed by 22F-inhibition ELISA. The reference cut-off value of the assay was an antibody concentration greater than or equal to (≥) 0.02 µg/mL.
Time Frame: At Month 3, one month after the administration of the third vaccine dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 185 | 177 | 183
Participants
  Anti-6A: number analyzed (Participants) | 185 | 176 | 183
  Anti-6A | 58 | 51 | 41
  Anti-19A: number analyzed (Participants) | 180 | 177 | 180
  Anti-19A | 56 | 50 | 40

6. Secondary Outcome: Antibody Concentrations Against Pneumococcal Cross-reactive Serotypes 6A and 19A (Anti-6A and 19A) - Primary Vaccination
Description: Anti-pneumococcal cross-reactive serotypes 6A and 19A antibody concentrations (Anti-6A and -19A) were measured by 22F-inhibition ELISA; presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (μg/mL). The seropositivity cut-off for the assay was ≥ 0.05 μg/mL.
Time Frame: At Month 3, one month after the administration of the third vaccine dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 185 | 177 | 183
µg/mL
  Anti-6A: number analyzed (Participants) | 185 | 176 | 183
  Anti-6A | 0.1 [0.08 to 0.12] | 0.1 [0.09 to 0.12] | 0.08 [0.06 to 0.09]
  Anti-19A: number analyzed (Participants) | 180 | 177 | 180
  Anti-19A | 0.1 [0.09 to 0.13] | 0.09 [0.08 to 0.11] | 0.08 [0.07 to 0.1]

7. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Cross-reactive Serotypes 6A and 19A - Primary Vaccination.
Description: Titers were presented as geometric mean titers (GMTs), for the seropositivity cut-off of 8.
Time Frame: At Month 3, one month after the administration of the third vaccine dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 135 | 129 | 130
Titers
  Opsono-6A: number analyzed (Participants) | 128 | 120 | 121
  Opsono-6A | 23.2 [16.1 to 33.6] | 25.4 [17.1 to 37.8] | 33 [21.4 to 50.8]
  Opsono-19A | 9 [6.9 to 11.7] | 8 [6.3 to 10.2] | 4.9 [4.4 to 5.4]

8. Secondary Outcome: Concentrations of Antibodies Against Diphtheria and Tetanus Toxoids (Anti-D and T) - Primary Vaccination
Description: Anti-D and anti-T antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in international units per milliliter (IU/mL). The seropositivity cut-off value was greater than or equal to (≥) 0.1 IU/mL.
Time Frame: At Month 3, one month after the administration of the third vaccine dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 187 | 180 | 189
IU/mL
  Anti-diphteria: number analyzed (Participants) | 185 | 176 | 187
  Anti-diphteria | 1.475 [1.307 to 1.664] | 1.078 [0.939 to 1.237] | 1.077 [0.949 to 1.222]
  Anti-tetanus | 2.873 [2.622 to 3.147] | 1.702 [1.528 to 1.897] | 0.934 [0.837 to 1.043]

9. Secondary Outcome: Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentrations - Primary Vaccination
Description: Anti-PRP antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (µg/mL). The seropositivity cut-off value was ≥ 0.15 µg/mL.
Time Frame: At Month 3, one month after the administration of the third vaccine dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 189 | 179 | 188
µg/mL | 2.139 [1.766 to 2.59] | 4.796 [3.829 to 6.007] | 2.219 [1.724 to 2.857]

10. Secondary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations - Primary Vaccination
Description: Anti-PT, anti-FHA and anti-PRN antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in ELISA units per milliliter (EL.U/mL). The seropositivity cut-off value was ≥ 5 EL.U/mL.
Time Frame: At Month 3, one month after the administration of the third vaccine dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 187 | 180 | 188
EL.U/mL
  Anti-PT | 42.7 [39.1 to 46.6] | 36.4 [33.4 to 39.8] | 40.1 [37 to 43.6]
  Anti-FHA: number analyzed (Participants) | 183 | 172 | 183
  Anti-FHA | 145.6 [130.4 to 162.5] | 100.8 [89.6 to 113.5] | 100.5 [89.9 to 112.4]
  Anti-PRN | 97.6 [86.8 to 109.7] | 40.1 [34.8 to 46.1] | 45.1 [39.3 to 51.7]

11. Secondary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations - Primary Vaccination.
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL). A seroprotected subject was a subject whose antibody ChemiLuminescence ImmunoAssay (CLIA) concentration was greater than or equal to the cut-off value ≥ 10 milli-international units per milliliter (mIU/mL). Note: investigations on the quality of some serology assays revealed that the anti-HBs ELISA overestimated concentration between 10-100 mIU/mL while values > 100 mIU/mL were confirmed valid. Therefore, all available samples at one month post-dose III and one month post-dose IV timepoints for which the anti-HBs antibody concentration was between 10-100 mIU/mL by in-house ELISA, were retested by the commercial assay Centaur™, an FDA-approved and CE-marked CLIA with a cut-off defining seropositivity of 6.2 mIU/mL. Anti-HBs seroprotection was redefined as in-house ELISA concentration > 100 mIU/mL or CLIA concentration > 10 mIU/mL.
Time Frame: At Month 3, one month after the administration of the third vaccine dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 111 | 112 | 113
mIU/mL | 356.9 [279.4 to 455.8] | 14 [11.6 to 16.9] | 11.5 [9.8 to 13.5]

12. Secondary Outcome: Anti-polio Types 1, 2 and 3 Titers - Primary Vaccination.
Description: Anti-polio 1, -polio 2, -polio 3 antibody titers were presented as geometric mean titers (GMTs), for the seropositivity cut-off value ≥ 8.
Time Frame: At Month 3, one month after the administration of the third vaccine dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 156 | 150 | 149
Titers
  Anti-polio 1: number analyzed (Participants) | 155 | 150 | 149
  Anti-polio 1 | 27.2 [21.7 to 34.1] | 16 [13 to 19.7] | 18.1 [14.8 to 22.1]
  Anti-polio 2: number analyzed (Participants) | 156 | 149 | 149
  Anti-polio 2 | 37.1 [29.1 to 47.4] | 29 [23 to 36.6] | 23.2 [18.5 to 29.1]
  Anti-polio 3: number analyzed (Participants) | 156 | 148 | 149
  Anti-polio 3 | 47.3 [35.8 to 62.4] | 34.2 [27 to 43.4] | 26.7 [21.5 to 33]

13. Secondary Outcome: Number of Subjects With Antibody Concentrations Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Anti-1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) ≥ 0.2 μg/mL - Booster Vaccination
Description: as for outcome 3
Time Frame: Prior to (Month 9) and one month after the administration of the booster dose (Month 10)
Population: The Booster ATP cohort for immunogenicity included all evaluable subjects, for whom assay results were available for antibodies against at least one study vaccine antigen component after booster vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 190 | 198 | 202
Participants
  Anti-1, Month 9: number analyzed (Participants) | 178 | 185 | 198
  Anti-1, Month 9 | 84 | 92 | 6
  Anti-4, Month 9: number analyzed (Participants) | 174 | 181 | 194
  Anti-4, Month 9 | 136 | 147 | 148
  Anti-5, Month 9: number analyzed (Participants) | 181 | 181 | 198
  Anti-5, Month 9 | 142 | 152 | 3
  Anti-6B, Month 9: number analyzed (Participants) | 175 | 180 | 192
  Anti-6B, Month 9 | 117 | 127 | 62
  Anti-7F, Month 9: number analyzed (Participants) | 176 | 181 | 195
  Anti-7F, Month 9 | 165 | 164 | 5
  Anti-9V, Month 9: number analyzed (Participants) | 180 | 180 | 196
  Anti-9V, Month 9 | 168 | 168 | 176
  Anti-14, Month 9: number analyzed (Participants) | 183 | 184 | 199
  Anti-14, Month 9 | 170 | 172 | 190
  Anti-18C, Month 9: number analyzed (Participants) | 179 | 181 | 194
  Anti-18C, Month 9 | 152 | 143 | 151
  Anti-19F, Month 9: number analyzed (Participants) | 172 | 177 | 197
  Anti-19F, Month 9 | 149 | 157 | 109
  Anti-23F, Month 9: number analyzed (Participants) | 180 | 182 | 196
  Anti-23F, Month 9 | 123 | 140 | 108
  Anti-1, Month 10: number analyzed (Participants) | 187 | 196 | 199
  Anti-1, Month 10 | 187 | 195 | 7
  Anti-4, Month 10: number analyzed (Participants) | 187 | 194 | 198
  Anti-4, Month 10 | 187 | 194 | 198
  Anti-5, Month 10: number analyzed (Participants) | 186 | 191 | 195
  Anti-5, Month 10 | 185 | 191 | 4
  Anti-6B, Month 10: number analyzed (Participants) | 186 | 193 | 199
  Anti-6B, Month 10 | 176 | 181 | 192
  Anti-7F, Month 10: number analyzed (Participants) | 189 | 198 | 199
  Anti-7F, Month 10 | 189 | 198 | 8
  Anti-9V, Month 10: number analyzed (Participants) | 188 | 197 | 202
  Anti-9V, Month 10 | 188 | 197 | 202
  Anti-14, Month 10: number analyzed (Participants) | 190 | 198 | 201
  Anti-14, Month 10 | 190 | 197 | 198
  Anti-18C, Month 10: number analyzed (Participants) | 189 | 197 | 200
  Anti-18C, Month 10 | 188 | 196 | 200
  Anti-19F, Month 10: number analyzed (Participants) | 183 | 194 | 196
  Anti-19F, Month 10 | 180 | 191 | 196
  Anti-23F, Month 10: number analyzed (Participants) | 185 | 194 | 199
  Anti-23F, Month 10 | 179 | 190 | 194

14. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Anti-1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) - Booster Vaccination
Description: Anti-pneumococcal serotype 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations were assessed by 22F-inhibition ELISA, presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (μg/mL). The seropositivity cut-off value was ≥ 0.05 μg/mL.
Time Frame: Prior (Month 9) to and one month after the administration of the booster dose (Month 10)
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 190 | 198 | 202
μg/mL
  Anti-1, Month 9: number analyzed (Participants) | 178 | 185 | 198
  Anti-1, Month 9 | 0.2 [0.17 to 0.22] | 0.22 [0.19 to 0.26] | 0.03 [0.03 to 0.04]
  Anti-4, Month 9: number analyzed (Participants) | 174 | 181 | 194
  Anti-4, Month 9 | 0.39 [0.34 to 0.46] | 0.43 [0.37 to 0.5] | 0.38 [0.34 to 0.43]
  Anti-5, Month 9: number analyzed (Participants) | 181 | 181 | 198
  Anti-5, Month 9 | 0.41 [0.36 to 0.47] | 0.42 [0.37 to 0.48] | 0.03 [0.03 to 0.04]
  Anti-6B, Month 9: number analyzed (Participants) | 175 | 180 | 192
  Anti-6B, Month 9 | 0.3 [0.25 to 0.36] | 0.32 [0.27 to 0.38] | 0.13 [0.11 to 0.16]
  Anti-7F, Month 9: number analyzed (Participants) | 176 | 181 | 195
  Anti-7F, Month 9 | 0.6 [0.54 to 0.68] | 0.62 [0.55 to 0.71] | 0.03 [0.03 to 0.03]
  Anti-9V, Month 9: number analyzed (Participants) | 180 | 180 | 196
  Anti-9V, Month 9 | 0.68 [0.6 to 0.78] | 0.76 [0.66 to 0.89] | 0.55 [0.49 to 0.62]
  Anti-14, Month 9: number analyzed (Participants) | 183 | 184 | 199
  Anti-14, Month 9 | 1.06 [0.9 to 1.26] | 1.14 [0.95 to 1.36] | 1.55 [1.35 to 1.79]
  Anti-18C, Month 9: number analyzed (Participants) | 179 | 181 | 194
  Anti-18C, Month 9 | 0.58 [0.49 to 0.68] | 0.43 [0.36 to 0.5] | 0.4 [0.35 to 0.45]
  Anti-19F, Month 9: number analyzed (Participants) | 172 | 177 | 197
  Anti-19F, Month 9 | 0.79 [0.64 to 0.99] | 0.9 [0.73 to 1.11] | 0.31 [0.25 to 0.37]
  Anti-23F, Month 9: number analyzed (Participants) | 180 | 182 | 196
  Anti-23F, Month 9 | 0.33 [0.27 to 0.39] | 0.38 [0.32 to 0.46] | 0.26 [0.22 to 0.3]
  Anti-1, Month 10: number analyzed (Participants) | 187 | 196 | 199
  Anti-1, Month 10 | 2.16 [1.89 to 2.46] | 2.5 [2.19 to 2.89] | 0.03 [0.03 to 0.04]
  Anti-4, Month 10: number analyzed (Participants) | 187 | 194 | 198
  Anti-4, Month 10 | 3.04 [2.7 to 3.42] | 3.29 [2.89 to 3.73] | 4.01 [3.53 to 4.56]
  Anti-5, Month 10: number analyzed (Participants) | 186 | 191 | 195
  Anti-5, Month 10 | 3.27 [2.9 to 3.7] | 3.27 [2.9 to 3.68] | 0.04 [0.03 to 0.04]
  Anti-6B, Month 10: number analyzed (Participants) | 186 | 193 | 199
  Anti-6B, Month 10 | 1.45 [1.23 to 1.71] | 1.41 [1.19 to 1.67] | 2.52 [2.15 to 2.96]
  Anti-7F, Month 10: number analyzed (Participants) | 189 | 198 | 199
  Anti-7F, Month 10 | 3.79 [3.4 to 4.23] | 4.06 [3.63 to 4.54] | 0.03 [0.03 to 0.04]
  Anti-9V, Month 10: number analyzed (Participants) | 188 | 197 | 202
  Anti-9V, Month 10 | 3.96 [3.58 to 4.39] | 4.23 [3.78 to 4.74] | 6.05 [5.38 to 6.8]
  Anti-14, Month 10: number analyzed (Participants) | 190 | 198 | 201
  Anti-14, Month 10 | 4.59 [4.06 to 5.19] | 4.95 [4.38 to 5.6] | 7.31 [6.37 to 8.39]
  Anti-18C, Month 10: number analyzed (Participants) | 189 | 197 | 200
  Anti-18C, Month 10 | 6.36 [5.56 to 7.27] | 4.63 [4.09 to 5.25] | 5.08 [4.47 to 5.78]
  Anti-19F, Month 10: number analyzed (Participants) | 183 | 194 | 196
  Anti-19F, Month 10 | 5.45 [4.72 to 6.3] | 5.8 [5.04 to 6.68] | 2.4 [2.14 to 2.7]
  Anti-23F, Month 10: number analyzed (Participants) | 185 | 194 | 199
  Anti-23F, Month 10 | 2.32 [1.98 to 2.71] | 2.6 [2.24 to 3.02] | 5.32 [4.49 to 6.31]

15. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F - Booster Vaccination
Description: Titers were presented as geometric mean titers (GMTs), for the seropositivity cut-off value of 8.
Time Frame: Prior (Month 9) to and one month after the administration of the booster dose(Month 10)
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 156 | 154 | 168
Titers
  Opsono-1, Month 9: number analyzed (Participants) | 149 | 152 | 168
  Opsono-1, Month 9 | 5.5 [4.7 to 6.4] | 5.6 [4.7 to 6.7] | 5 [4.4 to 5.8]
  Opsono-4, Month 9: number analyzed (Participants) | 145 | 150 | 164
  Opsono-4, Month 9 | 11.3 [8.6 to 14.9] | 15.3 [11.3 to 20.6] | 12.3 [9.3 to 16.2]
  Opsono-5, Month 9: number analyzed (Participants) | 148 | 151 | 166
  Opsono-5, Month 9 | 7.2 [6.1 to 8.5] | 7 [6 to 8.1] | 4.3 [4 to 4.6]
  Opsono-6B, Month 9: number analyzed (Participants) | 141 | 138 | 153
  Opsono-6B, Month 9 | 52 [34.8 to 77.7] | 96.7 [63.1 to 148] | 27.4 [18.6 to 40.3]
  Opsono-7F, Month 9: number analyzed (Participants) | 146 | 150 | 146
  Opsono-7F, Month 9 | 818.9 [642.2 to 1044.3] | 754.3 [598.4 to 950.8] | 138.1 [91.2 to 209.2]
  Opsono-9V, Month 9: number analyzed (Participants) | 143 | 147 | 159
  Opsono-9V, Month 9 | 267.2 [212.7 to 335.8] | 338.7 [264.8 to 433.2] | 149.5 [112.4 to 198.9]
  Opsono-14, Month 9: number analyzed (Participants) | 143 | 144 | 161
  Opsono-14, Month 9 | 117.3 [82.9 to 165.9] | 142.5 [101.3 to 200.4] | 156 [114.5 to 212.5]
  Opsono-18C, Month 9: number analyzed (Participants) | 139 | 148 | 162
  Opsono-18C, Month 9 | 8.2 [6.2 to 10.8] | 6.8 [5.3 to 8.5] | 7 [5.7 to 8.7]
  Opsono-19F, Month 9: number analyzed (Participants) | 149 | 149 | 167
  Opsono-19F, Month 9 | 13.8 [10.6 to 18.1] | 15.4 [11.8 to 20.2] | 7.8 [6.2 to 9.9]
  Opsono-23F, Month 9: number analyzed (Participants) | 143 | 143 | 162
  Opsono-23F, Month 9 | 314.1 [198.6 to 496.7] | 350.4 [229.8 to 534.2] | 338.9 [219.9 to 522.3]
  Opsono-1, Month 10: number analyzed (Participants) | 156 | 154 | 164
  Opsono-1, Month 10 | 208.8 [106.6 to 271.7] | 221.4 [165.1 to 297] | 4.6 [4.2 to 5.1]
  Opsono-4, Month 10: number analyzed (Participants) | 155 | 152 | 164
  Opsono-4, Month 10 | 1046.8 [865.8 to 1265.7] | 1121.6 [909.4 to 1383.3] | 2335.8 [1946.3 to 2803.3]
  Opsono-5, Month 10: number analyzed (Participants) | 152 | 151 | 164
  Opsono-5, Month 10 | 149.3 [119.2 to 187] | 132.4 [103.8 to 168.9] | 4.1 [4 to 4.3]
  Opsono-6B, Month 10: number analyzed (Participants) | 153 | 149 | 160
  Opsono-6B, Month 10 | 681.4 [514.6 to 902.1] | 763.3 [581.9 to 1001.3] | 1807.5 [1408 to 2320.3]
  Opsono-7F, Month 10: number analyzed (Participants) | 154 | 152 | 153
  Opsono-7F, Month 10 | 3936.5 [3413.2 to 4540] | 3976 [3390.2 to 4663.1] | 129.1 [85.9 to 193.9]
  Opsono-9V, Month 10: number analyzed (Participants) | 153 | 151 | 163
  Opsono-9V, Month 10 | 2512.9 [2213.1 to 2853.2] | 2257.6 [1974.3 to 2581.5] | 3889.5 [3260.1 to 4640.2]
  Opsono-14, Month 10: number analyzed (Participants) | 154 | 154 | 164
  Opsono-14, Month 10 | 1534.2 [1290.9 to 1823.3] | 1896.3 [1591.3 to 2259.7] | 1867.9 [1540.5 to 2265.1]
  Opsono-18C, Month 10: number analyzed (Participants) | 153 | 152 | 159
  Opsono-18C, Month 10 | 720.7 [597.5 to 869.4] | 385.9 [303.5 to 490.8] | 660.4 [520.9 to 837.3]
  Opsono-19F, Month 10: number analyzed (Participants) | 153 | 149 | 164
  Opsono-19F, Month 10 | 435.7 [336.3 to 564.5] | 475.4 [377.8 to 598.1] | 123.2 [95.9 to 158.2]
  Opsono-23F, Month 10: number analyzed (Participants) | 152 | 154 | 164
  Opsono-23F, Month 10 | 2895.4 [2276.1 to 3683.1] | 2895.3 [2419.3 to 3465] | 12418.7 [10171.8 to 15161.9]

16. Secondary Outcome: Number of Subjects With Antibody Concentrations Against Pneumococcal Cross-reactive Serotypes 6A and 19A (Anti-6A and 19A) ≥ 0.2 μg/mL - Booster Vaccination.
Description: Antibody concentrations against the cross-reactive pneumococcal serotypes were assessed by 22F-inhibition ELISA. The reference cut-off value of the assay was an antibody concentration greater than or equal to (≥) 0.02 µg/mL.
Time Frame: Prior (Month 9) to and one month after the administration of the booster dose(Month 10)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 187 | 196 | 201
Participants
  Anti-6A, Month 9: number analyzed (Participants) | 181 | 185 | 193
  Anti-6A, Month 9 | 50 | 56 | 28
  Anti-19A, Month 9: number analyzed (Participants) | 182 | 184 | 199
  Anti-19A, Month 9 | 61 | 63 | 29
  Anti-6A, Month 10 | 135 | 142 | 160
  Anti-19A, Month 10: number analyzed (Participants) | 187 | 195 | 200
  Anti-19A, Month 10 | 130 | 139 | 97

17. Secondary Outcome: Antibody Concentrations Against Pneumococcal Cross-reactive Serotypes 6A and 19A (Anti-6A and 19A) - Booster Vaccination
Description: Anti-pneumococcal cross-reactive serotype 6A and 19A antibody concentrations were assessed by 22F-inhibition ELISA, presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (μg/mL). The seropositivity cut-off value was ≥ 0.05 μg/mL.
Time Frame: Prior (Month 9) to and one month after the administration of the booster dose (Month 10)
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 187 | 196 | 201
μg/mL
  Anti-6A, Month 9: number analyzed (Participants) | 181 | 185 | 193
  Anti-6A, Month 9 | 0.1 [0.09 to 0.12] | 0.11 [0.09 to 0.13] | 0.06 [0.05 to 0.07]
  Anti-19A, Month 9: number analyzed (Participants) | 182 | 184 | 199
  Anti-19A, Month 9 | 0.12 [0.1 to 0.15] | 0.12 [0.09 to 0.13] | 0.06 [0.05 to 0.07]
  Anti-6A, Month 10 | 0.45 [0.36 to 0.55] | 0.49 [0.4 to 0.61] | 0.71 [0.58 to 0.88]
  Anti-19A, Month 10: number analyzed (Participants) | 187 | 195 | 200
  Anti-19A, Month 10 | 0.5 [0.39 to 0.63] | 0.52 [0.41 to 0.66] | 0.21 [0.17 to 0.25]

18. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Cross-reactive Serotypes 6A and 19A - Booster Vaccination.
Description: Titers were presented as geometric mean titers (GMTs), for the seropositivity cut-off value of 8.
Time Frame: Prior to (Month 9) and one month after the administration of the booster dose (Month 10)
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 151 | 148 | 167
Titers
  Opsono-6A, Month 9: number analyzed (Participants) | 128 | 135 | 151
  Opsono-6A, Month 9 | 23.3 [15.7 to 34.6] | 30.7 [20.8 to 45.2] | 15.5 [11.1 to 21.6]
  Opsono-19A, Month 9: number analyzed (Participants) | 148 | 148 | 167
  Opsono-19A, Month 9 | 5.7 [4.6 to 7] | 5.5 [4.6 to 6.5] | 5.5 [4.6 to 6.5]
  Opsono-6A, Month 10: number analyzed (Participants) | 145 | 142 | 160
  Opsono-6A, Month 10 | 143.3 [99.1 to 207.3] | 197.1 [138 to 281.3] | 493.3 [357.1 to 681.6]
  Opsono-19A, Month 10: number analyzed (Participants) | 151 | 148 | 162
  Opsono-19A, Month 10 | 34.9 [24.8 to 49.2] | 24.6 [17.7 to 34.3] | 7.7 [6.2 to 9.5]

19. Secondary Outcome: Concentrations of Antibodies Against Protein D (Anti-PD) - Booster Vaccination.
Description: as for outcome 2
Time Frame: Prior (Month 9) to and one month after (Month 10) the administration of the booster dose
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 189 | 198 | 201
EL.U/mL
  Anti-PD, Month 9: number analyzed (Participants) | 182 | 189 | 195
  Anti-PD, Month 9 | 421 [370.3 to 478.5] | 520.5 [455.8 to 594.3] | 80.8 [73.1 to 89.4]
  Anti-PD, Month 10 | 1715 [1510.3 to 1947.5] | 1936.8 [1710.5 to 2193.2] | 84.1 [76 to 93.1]

20. Secondary Outcome: Concentrations of Antibodies Against Diphtheria and Tetanus Toxoids (Anti-D and T) - Booster Vaccination.
Description: as for outcome 8
Time Frame: Prior to (Month 9) and one month after (Month 10) the administration of the booster dose
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 186 | 194 | 197
IU/mL
  Anti-diphteria, Month 9: number analyzed (Participants) | 175 | 179 | 192
  Anti-diphteria, Month 9 | 0.235 [0.205 to 0.27] | 0.232 [0.203 to 0.264] | 0.266 [0.235 to 0.301]
  Anti-tetanus, Month 9: number analyzed (Participants) | 175 | 180 | 193
  Anti-tetanus, Month 9 | 0.728 [0.656 to 0.809] | 0.536 [0.477 to 0.603] | 0.232 [0.202 to 0.267]
  Anti-diphteria, Month 10 | 4.061 [3.601 to 4.58] | 3.226 [2.866 to 3.632] | 4.882 [4.425 to 5.386]
  Anti-tetanus, Month 10 | 8.628 [7.867 to 9.462] | 5.989 [5.461 to 6.568] | 3.248 [2.859 to 3.69]

21. Secondary Outcome: Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentrations - Booster Vaccination
Description: as for outcome 9
Time Frame: Prior to (Month 9) and one month after (Month 10) the administration of the booster dose
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 184 | 192 | 197
µg/mL
  Anti-PRP, Month 9: number analyzed (Participants) | 174 | 179 | 193
  Anti-PRP, Month 9 | 0.475 [0.386 to 0.585] | 0.855 [0.682 to 1.072] | 0.371 [0.298 to 0.461]
  Anti-PRP, Month 10 | 19.331 [16.144 to 23.147] | 39.383 [32.617 to 47.551] | 23.676 [18.944 to 29.591]

22. Secondary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations - Booster Vaccination.
Description: as for outcome 10
Time Frame: Prior (Month 9) to and one month after (Month 10) the administration of the booster dose
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 186 | 194 | 197
EL.U/mL
  Anti-PT, Month 9: number analyzed (Participants) | 174 | 176 | 189
  Anti-PT, Month 9 | 7.4 [6.6 to 8.4] | 6 [5.4 to 6.7] | 6.6 [5.9 to 7.3]
  Anti-FHA, Month 9: number analyzed (Participants) | 175 | 179 | 191
  Anti-FHA, Month 9 | 34 [29.4 to 39.4] | 35.3 [30.8 to 40.6] | 34.7 [30.1 to 39.9]
  Anti-PRN, Month 9: number analyzed (Participants) | 175 | 179 | 192
  Anti-PRN, Month 9 | 14.1 [12.3 to 16.2] | 6.8 [5.9 to 7.9] | 8.6 [7.4 to 10]
  Anti-PT, Month 10: number analyzed (Participants) | 186 | 194 | 196
  Anti-PT, Month 10 | 53.5 [48.3 to 59.2] | 47.4 [42.9 to 52.5] | 54.8 [48.9 to 61.4]
  Anti-FHA, Month 10: number analyzed (Participants) | 184 | 192 | 194
  Anti-FHA, Month 10 | 343.5 [308 to 383.1] | 135.7 [121.2 to 151.9] | 140 [123.2 to 159.1]
  Anti-PRN, Month 10: number analyzed (Participants) | 186 | 193 | 197
  Anti-PRN, Month 10 | 281.7 [247.2 to 321] | 97.8 [85.4 to 112] | 106.4 [91.5 to 123.8]

23. Secondary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations - Booster Vaccination.
Description: as for outcome 11
Time Frame: Prior (Month 9) to and one month after (Month 10) the administration of the booster dose
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 125 | 124 | 135
mIU/mL
  Anti-HBs, Month 9: number analyzed (Participants) | 121 | 124 | 135
  Anti-HBs, Month 9 | 142.1 [113.4 to 178.1] | 9.9 [8.8 to 11.2] | 9.9 [8.8 to 11.2]
  Anti-HBs, Month 10: number analyzed (Participants) | 125 | 123 | 135
  Anti-HBs, Month 10 | 1981 [1552 to 2528.7] | 8.6 [7.6 to 9.9] | 8.5 [7.6 to 9.5]

24. Secondary Outcome: Anti-polio Types 1, 2 and 3 Titers - Booster Vaccination.
Description: as for outcome 12
Time Frame: Prior (Month 9) to and one month after (Month 10) the administration of the booster dose
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 167 | 173 | 182
Titers
  Anti-polio 1, Month 9: number analyzed (Participants) | 156 | 166 | 182
  Anti-polio 1, Month 9 | 8.3 [7 to 10] | 7.3 [6.3 to 8.4] | 7 [6.1 to 8]
  Anti-polio 2, Month 9: number analyzed (Participants) | 156 | 164 | 182
  Anti-polio 2, Month 9 | 13.4 [10.8 to 16.6] | 10.6 [8.8 to 12.7] | 10.4 [8.9 to 12.2]
  Anti-polio 3, Month 9: number analyzed (Participants) | 156 | 166 | 180
  Anti-polio 3, Month 9 | 11.3 [9.3 to 13.9] | 9 [7.5 to 10.7] | 8.7 [7.4 to 10.3]
  Anti-polio 1, Month 10: number analyzed (Participants) | 166 | 173 | 170
  Anti-polio 1, Month 10 | 370.7 [289.8 to 474.2] | 177.5 [135.8 to 231.9] | 221.2 [171.5 to 285.3]
  Anti-polio 2, Month 10: number analyzed (Participants) | 167 | 173 | 169
  Anti-polio 2, Month 10 | 710.8 [588 to 859] | 338.8 [272.7 to 420.8] | 481.4 [391 to 592.7]
  Anti-polio 3, Month 10: number analyzed (Participants) | 167 | 172 | 170
  Anti-polio 3, Month 10 | 631.5 [495.7 to 804.4] | 311.9 [240.4 to 404.6] | 348.3 [263.6 to 460.2]

25. Secondary Outcome: Number of Subjects With Booster Vaccine Response Against Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN) Antibodies - Booster Vaccination.
Description: A booster responder to PT/FHA/PRN was defined as a subject with antibodies concentration ≥ 5 EL.U/mL against PT/FHA/PRN in subjects who were initially seronegative for anti-PT/FHA/PRN antibodies (i.e., subjects with anti-PT/FHA/PRN antibody concentrations < 5 EL.U/mL), or antibody concentration ≥ 2 fold the pre-vaccination antibody concentration in subjects who were initially seropositive (i.e., subjects with anti-PT/FHA/PRN antibody concentrations ≥ 5 EL.U/mL).
Time Frame: One month after (Month 10) the administration of the booster dose
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 140 | 145 | 155
Participants
  Anti-PT, S- seronegative: number analyzed (Participants) | 40 | 48 | 48
  Anti-PT, S- seronegative | 40 | 47 | 48
  Anti-PT, S+ seropositive: number analyzed (Participants) | 99 | 95 | 105
  Anti-PT, S+ seropositive | 95 | 94 | 98
  Anti-FHA, S- seronegative: number analyzed (Participants) | 4 | 1 | 2
  Anti-FHA, S- seronegative | 4 | 1 | 2
  Anti-FHA, S+ seropositive: number analyzed (Participants) | 135 | 143 | 150
  Anti-FHA, S+ seropositive | 128 | 119 | 125
  Anti-PRN, S- seronegative: number analyzed (Participants) | 18 | 56 | 53
  Anti-PRN, S- seronegative | 18 | 56 | 51
  Anti-PRN, S+ seropositive: number analyzed (Participants) | 122 | 89 | 102
  Anti-PRN, S+ seropositive | 122 | 88 | 101

26. Secondary Outcome: Number of Subjects With Antibody Concentrations Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Anti-1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) ≥ 0.2 μg/mL - 12 Months After Booster Dose.
Description: as for outcome 3
Time Frame: At Month 21, 12 months after the administration of the booster dose (at 23-25 months of age)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 166 | 169 | 177
Participants
  Anti-1, Month 21: number analyzed (Participants) | 163 | 166 | 173
  Anti-1, Month 21 | 106 | 108 | 6
  Anti-4, Month 21: number analyzed (Participants) | 163 | 167 | 173
  Anti-4, Month 21 | 101 | 102 | 130
  Anti-5, Month 21: number analyzed (Participants) | 163 | 163 | 170
  Anti-5, Month 21 | 129 | 129 | 10
  Anti-6B, Month 21: number analyzed (Participants) | 162 | 164 | 173
  Anti-6B, Month 21 | 94 | 96 | 133
  Anti-7F, Month 21: number analyzed (Participants) | 163 | 165 | 170
  Anti-7F, Month 21 | 157 | 157 | 15
  Anti-9V, Month 21: number analyzed (Participants) | 165 | 168 | 173
  Anti-9V, Month 21 | 155 | 157 | 160
  Anti-14, Month 21 | 149 | 156 | 173
  Anti-18C, Month 21: number analyzed (Participants) | 164 | 167 | 174
  Anti-18C, Month 21 | 160 | 155 | 161
  Anti-19F, Month 21: number analyzed (Participants) | 164 | 165 | 171
  Anti-19F, Month 21 | 158 | 158 | 134
  Anti-23F, Month 21: number analyzed (Participants) | 162 | 166 | 172
  Anti-23F, Month 21 | 123 | 126 | 153

27. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Anti-1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) - 12 Months After Booster Dose.
Description: as for outcome 14
Time Frame: At Month 21, 12 months after the administration of the booster dose (at 23-25 months of age)
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 166 | 169 | 177
μg/mL
  Anti-1, Month 21: number analyzed (Participants) | 163 | 166 | 173
  Anti-1, Month 21 | 0.3 [0.26 to 0.35] | 0.32 [0.28 to 0.38] | 0.04 [0.03 to 0.04]
  Anti-4, Month 21: number analyzed (Participants) | 163 | 167 | 173
  Anti-4, Month 21 | 0.25 [0.22 to 0.29] | 0.29 [0.25 to 0.34] | 0.36 [0.32 to 0.42]
  Anti-5, Month 21: number analyzed (Participants) | 163 | 163 | 170
  Anti-5, Month 21 | 0.45 [0.39 to 0.53] | 0.47 [0.39 to 0.55] | 0.05 [0.04 to 0.05]
  Anti-6B, Month 21: number analyzed (Participants) | 162 | 164 | 173
  Anti-6B, Month 21 | 0.3 [0.25 to 0.36] | 0.32 [0.26 to 0.4] | 0.46 [0.38 to 0.56]
  Anti-7F, Month 21: number analyzed (Participants) | 163 | 165 | 170
  Anti-7F, Month 21 | 0.72 [0.63 to 0.81] | 0.73 [0.64 to 0.84] | 0.04 [0.03 to 0.05]
  Anti-9V, Month 21: number analyzed (Participants) | 165 | 168 | 173
  Anti-9V, Month 21 | 0.74 [0.63 to 0.88] | 0.78 [0.66 to 0.91] | 0.81 [0.7 to 0.94]
  Anti-14, Month 21 | 0.73 [0.62 to 0.86] | 0.85 [0.73 to 0.99] | 1.28 [1.1 to 1.48]
  Anti-18C, Month 21: number analyzed (Participants) | 164 | 167 | 174
  Anti-18C, Month 21 | 1.03 [0.89 to 1.19] | 0.64 [0.56 to 0.74] | 1.66 [1.59 to 1.75]
  Anti-19F, Month 21: number analyzed (Participants) | 164 | 165 | 171
  Anti-19F, Month 21 | 1.48 [1.22 to 1.8] | 1.46 [1.2 to 1.78] | 1.76 [1.59 to 1.98]
  Anti-23F, Month 21: number analyzed (Participants) | 162 | 166 | 172
  Anti-23F, Month 21 | 0.51 [0.41 to 0.63] | 0.52 [0.42 to 1.63] | 1.01 [0.83 to 1.24]

28. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F - 12 Months After Booster Dose.
Description: Titers were presented as geometric mean titers (GMTs), for the seropositivity cut-off value of 8.
Time Frame: At Month 21, 12 months after the administration of the booster dose (at 23-25 months of age)
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 159 | 152 | 165
Titers
  Opsono-1, Month 21: number analyzed (Participants) | 159 | 150 | 162
  Opsono-1, Month 21 | 10.9 [8.5 to 14.1] | 9.9 [7.8 to 12.5] | 4.3 [3.9 to 4.7]
  Opsono-4, Month 21: number analyzed (Participants) | 154 | 147 | 160
  Opsono-4, Month 21 | 12 [9.1 to 15.9] | 15.5 [11 to 21.7] | 45.2 [30.8 to 66.5]
  Opsono-5, Month 21 | 12.9 [10.4 to 16] | 13.7 [11 to 17.1] | 4.1 [3.9 to 4.3]
  Opsono-6B, Month 21: number analyzed (Participants) | 139 | 137 | 152
  Opsono-6B, Month 21 | 77.7 [48.8 to 123.8] | 137.6 [83.5 to 226.6] | 220 [145.4 to 332.8]
  Opsono-7F, Month 21: number analyzed (Participants) | 142 | 136 | 143
  Opsono-7F, Month 21 | 1982.9 [1568.8 to 2506.2] | 2205.6 [1833.4 to 2653.4] | 738.1 [549.8 to 990.7]
  Opsono-9V, Month 21: number analyzed (Participants) | 143 | 135 | 147
  Opsono-9V, Month 21 | 465.9 [324.2 to 669.5] | 470 [325.8 to 677.9] | 476.2 [317.8 to 713.5]
  Opsono-14, Month 21: number analyzed (Participants) | 128 | 121 | 149
  Opsono-14, Month 21 | 93.1 [60 to 144.4] | 151.6 [97.7 to 235.4] | 238.7 [163.5 to 348.6]
  Opsono-18C, Month 21: number analyzed (Participants) | 135 | 133 | 151
  Opsono-18C, Month 21 | 21.6 [15.2 to 30.6] | 12.5 [8.9 to 17.6] | 15.3 [10.9 to 21.3]
  Opsono-19F, Month 21: number analyzed (Participants) | 148 | 150 | 162
  Opsono-19F, Month 21 | 31.1 [22.6 to 42.8] | 32.9 [23.8 to 45.4] | 15.1 [11 to 20.6]
  Opsono-23F, Month 21: number analyzed (Participants) | 146 | 140 | 161
  Opsono-23F, Month 21 | 366.5 [218.3 to 615.3] | 706.1 [443.5 to 1124.3] | 3879.8 [2774.4 to 5425.5]

29. Secondary Outcome: Number of Subjects With Antibody Concentrations Against Pneumococcal Cross-reactive Serotypes 6A and 19A (Anti-6A and 19A) ≥ 0.2 μg/mL - 12 Months After Booster Dose.
Description: as for outcome 16
Time Frame: At Month 21, 12 months after the administration of the booster dose (at 23-25 months of age)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 165 | 166 | 176
Participants
  Anti-6A, Month 21: number analyzed (Participants) | 163 | 166 | 174
  Anti-6A, Month 21 | 54 | 57 | 92
  Anti-19A, Month 21 | 120 | 97 | 80

30. Secondary Outcome: Antibody Concentrations Against Pneumococcal Cross-reactive Serotypes 6A and 19A (Anti-6A and 19A) - 12 Months After Booster Dose.
Description: as for outcome 17
Time Frame: At Month 21, 12 months after the administration of the booster dose (at 23-25 months of age)
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 165 | 166 | 176
μg/mL
  Anti-6A, Month 21: number analyzed (Participants) | 163 | 166 | 174
  Anti-6A, Month 21 | 0.14 [0.12 to 0.17] | 0.15 [0.12 to 0.19] | 0.22 [0.18 to 0.27]
  Anti-19A, Month 21 | 0.43 [0.35 to 0.53] | 0.29 [0.23 to 0.36] | 0.21 [0.16 to 0.27]

31. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Cross-reactive Serotypes 6A and 19A - 12 Months After Booster Dose.
Description: Titers were presented as geometric mean titers (GMTs), for the seropositivity cut-off value of 8.
Time Frame: At Month 21, 12 months after the administration of the booster dose (at 23-25 months of age)
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 150 | 146 | 158
Titers
  Opsono-6A, Month 21: number analyzed (Participants) | 126 | 129 | 148
  Opsono-6A, Month 21 | 21.6 [14.1 to 33.1] | 24.8 [15.5 to 39.5] | 56.5 [36.4 to 87.7]
  Opsono-19A, Month 21 | 12.6 [9.5 to 16.7] | 9.1 [7 to 11.9] | 9.6 [7.1 to 12.9]

32. Secondary Outcome: Concentrations of Antibodies Against Protein D (Anti-PD) - 12 Months After Booster Dose.
Description: as for outcome 2
Time Frame: At Month 21, 12 months after the administration of the booster dose (at 23-25 months of age)
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 168 | 170 | 178
EL.U/mL | 332 [287.1 to 384] | 423 [359.9 to 497.1] | 81.4 [73.1 to 90.6]

33. Secondary Outcome: Number of Subjects With Positive Cultures of Haemophilus Influenzae and/or Streptococcus Pneumoniae in the Nasopharynx - Primary Vaccination.
Description: Positive cultures of H. influenzae* (HI) and S. pneumoniae (SP) identified in the nasopharynx at each swab time point: one month post-Dose III (M3), M9 (11-13 months of age), M12 (14-16 months of age), M16 (18-20 months of age) and M21 (23-25 months of age). *Data presented only include results from samples confirmed as positive for H. influenzae / Non-typeable H. influenzae after differentiation from H. haemolyticus by Polymerase Chain Reaction (PCR) assay.
Time Frame: One month after the third dose (Month 3), prior to the booster dose (Month 9), 3 months after the booster dose (Month 12), 7 months after the booster dose (Month 16) and 12 months after the booster dose (Month 21)
Population: The Primary Total Vaccinated cohort included all vaccinated subjects who received at least one primary dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 260 | 259 | 259
Participants
  Any SP, Month 3 | 102 | 109 | 100
  Any SP, Month 9: number analyzed (Participants) | 255 | 259 | 258
  Any SP, Month 9 | 115 | 134 | 119
  Any SP, Month 12: number analyzed (Participants) | 256 | 258 | 257
  Any SP, Month 12 | 121 | 131 | 126
  Any SP, Month 16: number analyzed (Participants) | 256 | 258 | 258
  Any SP, Month 16 | 151 | 135 | 148
  Any SP, Month 21: number analyzed (Participants) | 255 | 257 | 257
  Any SP, Month 21 | 154 | 139 | 131
  Any HI, Month 3: number analyzed (Participants) | 259 | 258 | 258
  Any HI, Month 3 | 94 | 91 | 85
  Any HI, Month 9: number analyzed (Participants) | 254 | 258 | 256
  Any HI, Month 9 | 152 | 155 | 144
  Any HI, Month 12: number analyzed (Participants) | 260 | 258 | 257
  Any HI, Month 12 | 159 | 160 | 165
  Any HI, Month 16: number analyzed (Participants) | 252 | 258 | 256
  Any HI, Month 16 | 185 | 169 | 162
  Any HI, Month 21: number analyzed (Participants) | 254 | 255 | 254
  Any HI, Month 21 | 192 | 192 | 177

34. Secondary Outcome: Number of Subjects With Positive Cultures of Streptococcus Pneumoniae Vaccine Seroptypes (VS), Cross-reactive Serotypes (CRS) or Other Serotypes (OS) in the Nasopharynx - Primary Vaccination.
Description: Positive cultures of S. pneumoniae (SP) identified in the nasopharynx at each swab time point: one month post-Dose III (M3), pre-booster vaccination (11-13 months of age), M12 (14-16 months of age), M16 (18-20 months of age) and M21 (23-25 months of age).
Time Frame: as for outcome 33
Population: The Primary Total Vaccinated cohort included all vaccinated subjects who received at least one primary dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 260 | 259 | 259
Participants
  S. pneumoniae, VS - M3 | 18 | 25 | 21
  S. pneumoniae, VS - M9: number analyzed (Participants) | 255 | 259 | 257
  S. pneumoniae, VS - M9 | 16 | 20 | 18
  S. pneumoniae, VS - M12: number analyzed (Participants) | 256 | 258 | 257
  S. pneumoniae, VS - M12 | 11 | 18 | 13
  S. pneumoniae, VS - M16: number analyzed (Participants) | 256 | 258 | 258
  S. pneumoniae, VS - M16 | 15 | 12 | 12
  S. pneumoniae, VS - M21: number analyzed (Participants) | 255 | 257 | 257
  S. pneumoniae, VS - M21 | 8 | 8 | 8
  S. pneumoniae, CRS - M3 | 25 | 32 | 20
  S. pneumoniae, CRS - M9: number analyzed (Participants) | 255 | 259 | 257
  S. pneumoniae, CRS - M9 | 15 | 30 | 25
  S. pneumoniae, CRS - M12: number analyzed (Participants) | 256 | 258 | 257
  S. pneumoniae, CRS - M12 | 25 | 26 | 27
  S. pneumoniae, CRS - M16: number analyzed (Participants) | 256 | 258 | 258
  S. pneumoniae, CRS - M16 | 33 | 33 | 31
  S. pneumoniae, CRS - M21: number analyzed (Participants) | 255 | 257 | 257
  S. pneumoniae, CRS - M21 | 28 | 13 | 25
  S. pneumoniae, OS - M3 | 45 | 40 | 51
  S. pneumoniae, OS - M9: number analyzed (Participants) | 255 | 259 | 257
  S. pneumoniae, OS - M9 | 69 | 61 | 60
  S. pneumoniae, OS - M12: number analyzed (Participants) | 256 | 258 | 257
  S. pneumoniae, OS - M12 | 74 | 69 | 70
  S. pneumoniae, OS - M16: number analyzed (Participants) | 256 | 258 | 258
  S. pneumoniae, OS - M16 | 86 | 67 | 89
  S. pneumoniae, OS - M21: number analyzed (Participants) | 255 | 257 | 257
  S. pneumoniae, OS - M21 | 97 | 81 | 80

35. Secondary Outcome: Number of Subjects With Acquisition of New Streptococcus Pneumoniae and Haemophilus Influenzae Strains Identified in Nasopharyngeal Swabs - Primary Vaccination.
Description: Acquisition of new H. influenzae* (HI) and S. pneumoniae (SP) strains, identified in the nasopharynx at each swab time point: pre-booster vaccination (11-13 months of age), M12 (14-16 months of age), M16 (18-20 months of age) and M21 (23-25 months of age). *Data presented only include results from samples confirmed as positive for H. influenzae / Non-typeable H. influenzae after differentiation from H. haemolyticus by Polymerase Chain Reaction (PCR) assay.
Time Frame: Prior to the booster dose (Month 9), 3 months after the booster dose (Month 12), 7 months after the booster dose (Month 16) and 12 months after the booster dose (Month 21)
Population: The Primary Total Vaccinated cohort included all vaccinated subjects who received at least one primary dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 256 | 259 | 258
Participants
  Any SP, M9: number analyzed (Participants) | 255 | 259 | 258
  Any SP, M9 | 103 | 114 | 107
  Any SP, M12: number analyzed (Participants) | 256 | 258 | 257
  Any SP, M12 | 86 | 95 | 90
  Any SP, M16: number analyzed (Participants) | 256 | 258 | 258
  Any SP, M16 | 128 | 105 | 125
  Any SP, M21: number analyzed (Participants) | 255 | 257 | 257
  Any SP, M21 | 132 | 113 | 110
  Any HI, M9: number analyzed (Participants) | 254 | 258 | 256
  Any HI, M9 | 88 | 84 | 83
  Any HI, M12: number analyzed (Participants) | 256 | 258 | 257
  Any HI, M12 | 47 | 48 | 58
  Any HI, M16: number analyzed (Participants) | 252 | 258 | 256
  Any HI, M16 | 71 | 55 | 64
  Any HI, M21: number analyzed (Participants) | 254 | 255 | 254
  Any HI, M21 | 73 | 75 | 71

36. Secondary Outcome: Number of Subjects With Acquisition of New Streptococcus Pneumoniae Vaccine Serotypes (VS), Cross-reactive Serotypes (CRS) or Other Serotypes (OS) Identified in Nasopharyngeal Swabs - Primary Vaccination.
Description: Acquisition of new S. pneumonia (SP) strains, identified in the nasopharynx at each swab time point: pre-booster vaccination (11-13 months of age), M12 (14-16 months of age), M16 (18-20 months of age) and M21 (23-25 months of age).
Time Frame: as for outcome 35
Population: The Primary Total Vaccinated cohort included all vaccinated subjects who received at least one primary dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 256 | 259 | 258
Participants
  S. pneumoniae, VS - M9: number analyzed (Participants) | 255 | 259 | 257
  S. pneumoniae, VS - M9 | 14 | 11 | 15
  S. pneumoniae, VS - M12: number analyzed (Participants) | 256 | 258 | 257
  S. pneumoniae, VS - M12 | 8 | 9 | 8
  S. pneumoniae, VS - M16: number analyzed (Participants) | 256 | 258 | 258
  S. pneumoniae, VS - M16 | 13 | 7 | 9
  S. pneumoniae, VS - M21: number analyzed (Participants) | 255 | 257 | 257
  S. pneumoniae, VS - M21 | 4 | 7 | 6
  S. pneumoniae, CRS - M9: number analyzed (Participants) | 255 | 259 | 257
  S. pneumoniae, CRS - M9 | 13 | 26 | 20
  S. pneumoniae, CRS - M12: number analyzed (Participants) | 256 | 258 | 257
  S. pneumoniae, CRS - M12 | 19 | 15 | 20
  S. pneumoniae, CRS - M16: number analyzed (Participants) | 256 | 258 | 258
  S. pneumoniae, CRS - M16 | 27 | 25 | 24
  S. pneumoniae, CRS - M21: number analyzed (Participants) | 255 | 257 | 257
  S. pneumoniae, CRS - M21 | 22 | 8 | 18
  S. pneumoniae, OS - M9: number analyzed (Participants) | 255 | 259 | 257
  S. pneumoniae, OS - M9 | 64 | 55 | 57
  S. pneumoniae, OS - M12: number analyzed (Participants) | 256 | 258 | 257
  S. pneumoniae, OS - M12 | 52 | 59 | 52
  S. pneumoniae, OS - M16: number analyzed (Participants) | 256 | 258 | 258
  S. pneumoniae, OS - M16 | 74 | 55 | 77
  S. pneumoniae, OS - M21: number analyzed (Participants) | 255 | 257 | 257
  S. pneumoniae, OS - M21 | 87 | 69 | 69

37. Secondary Outcome: Number of Subjects With Solicited Local Symptoms - Primary Vaccination
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any occurrence of the specified symptom regardless of intensity. Grade 3 pain was defined as cried when limb was moved/spontaneously painful. Grade 3 redness/swelling was defined as redness/swelling spreading beyond (>) 30 millimeters from injection site.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each dose and across doses
Population: The Primary Total Vaccinated cohort included all vaccinated subjects who received at least one primary dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 260 | 260 | 260
Participants
  Any Pain, Dose 1 | 168 | 159 | 142
  Grade 3 Pain, Dose 1 | 30 | 31 | 22
  Any Redness, Dose 1 | 105 | 134 | 120
  Grade 3 Redness, Dose 1 | 7 | 21 | 15
  Any Swelling, Dose 1 | 140 | 145 | 113
  Grade 3 Swelling, Dose 1 | 12 | 18 | 15
  Any Pain, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Any Pain, Dose 2 | 130 | 120 | 104
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Grade 3 Pain, Dose 2 | 11 | 12 | 13
  Any Redness, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Any Redness, Dose 2 | 125 | 131 | 121
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Grade 3 Redness, Dose 2 | 4 | 8 | 4
  Any Swelling, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Any Swelling, Dose 2 | 143 | 135 | 125
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Grade 3 Swelling, Dose 2 | 7 | 8 | 8
  Any Pain, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Any Pain, Dose 3 | 100 | 87 | 73
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Grade 3 Pain, Dose 3 | 9 | 4 | 5
  Any Redness, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Any Redness, Dose 3 | 141 | 119 | 121
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Grade 3 Redness, Dose 3 | 1 | 1 | 1
  Any Swelling, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Any Swelling, Dose 3 | 142 | 133 | 118
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Grade 3 Swelling, Dose 3 | 4 | 7 | 10
  Any Pain, Across doses | 205 | 193 | 178
  Grade 3 Pain, Across doses | 42 | 40 | 29
  Any Redness, Across doses | 197 | 193 | 184
  Grade 3 Redness, Across doses | 12 | 26 | 19
  Any Swelling, Across doses | 205 | 199 | 179
  Grade 3 Swelling, Across doses | 18 | 29 | 24

38. Secondary Outcome: Number of Subjects With Solicited General Symptoms - Primary Vaccination
Description: Solicited general symptoms assessed include drowsiness, fever (defined as rectal temperature ≥ 38.0°C), irritability, and loss of appetite. Any was defined as incidence of the specified symptom regardless of intensity. Grade 3 drowsiness was defined as drowsiness which prevented normal everyday activities. Grade 3 fever was defined as fever (rectal temperature) above (>) 40.0 degree Celsius (°C). Grade 3 irritability was defined as crying that could not be comforted/preventing normal activity. Grade 3 loss of appetite was defined as the subject not eating at all. Related symptom was defined as a general symptom assessed by the investigator as causally related to study vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each dose and across doses
Population: The Primary Total Vaccinated cohort included all vaccinated subjects who received at least one primary dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 260 | 260 | 260
Participants
  Any Drowsiness, Dose 1 | 183 | 171 | 164
  Grade 3 Drowsiness, Dose 1 | 4 | 7 | 6
  Related Drowsiness, Dose 1 | 178 | 171 | 160
  Any Temperature, Dose 1 | 88 | 63 | 40
  Grade 3 Temperature, Dose 1 | 0 | 0 | 0
  Related Temperature, Dose 1 | 88 | 62 | 40
  Any Irritability, Dose 1 | 190 | 185 | 180
  Grade 3 Irritability, Dose 1 | 18 | 18 | 8
  Related Irritability, Dose 1 | 186 | 182 | 173
  Any Loss of appetite, Dose 1 | 88 | 94 | 87
  Grade 3 Loss of appetite, Dose 1 | 3 | 0 | 1
  Related Loss of appetite, Dose 1 | 85 | 94 | 84
  Any Drowsiness, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Any Drowsiness, Dose 2 | 157 | 141 | 143
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Grade 3 Drowsiness, Dose 2 | 5 | 5 | 1
  Related Drowsiness, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Related Drowsiness, Dose 2 | 152 | 141 | 141
  Any Temperature, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Any Temperature, Dose 2 | 82 | 60 | 60
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Grade 3 Temperature, Dose 2 | 0 | 0 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Related Temperature, Dose 2 | 81 | 58 | 59
  Any Irritability, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Any Irritability, Dose 2 | 181 | 176 | 165
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Grade 3 Irritability, Dose 2 | 14 | 12 | 5
  Related Irritability, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Related Irritability, Dose 2 | 177 | 172 | 154
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Any Loss of appetite, Dose 2 | 82 | 73 | 85
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Grade 3 Loss of appetite, Dose 2 | 1 | 2 | 0
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 259 | 260 | 260
  Related Loss of appetite, Dose 2 | 80 | 69 | 81
  Any Drowsiness, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Any Drowsiness, Dose 3 | 127 | 114 | 118
  Grade 3 Drowsiness, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Grade 3 Drowsiness, Dose 3 | 7 | 3 | 1
  Related Drowsiness, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Related Drowsiness, Dose 3 | 124 | 111 | 115
  Any Temperature, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Any Temperature, Dose 3 | 70 | 50 | 38
  Grade 3 Temperature, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Grade 3 Temperature, Dose 3 | 0 | 0 | 0
  Related Temperature, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Related Temperature, Dose 3 | 67 | 47 | 34
  Any Irritability, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Any Irritability, Dose 3 | 138 | 137 | 138
  Grade 3 Irritability, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Grade 3 Irritability, Dose 3 | 19 | 15 | 5
  Related Irritability, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Related Irritability, Dose 3 | 132 | 133 | 133
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Any Loss of appetite, Dose 3 | 63 | 59 | 59
  Grade 3 Loss of appetite, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Grade 3 Loss of appetite, Dose 3 | 0 | 2 | 0
  Related Loss of appetite, Dose 3: number analyzed (Participants) | 260 | 259 | 260
  Related Loss of appetite, Dose 3 | 58 | 55 | 54
  Any Drowsiness, Across doses | 231 | 220 | 215
  Grade 3 Drowsiness, Across doses | 14 | 13 | 7
  Related Drowsiness, Across doses | 227 | 219 | 213
  Any Temperature, Across doses | 153 | 124 | 110
  Grade 3 Temperature, Across doses | 0 | 0 | 0
  Related Temperature, Across doses | 149 | 120 | 106
  Any Irritability, Across doses | 241 | 230 | 235
  Grade 3 Irritability, Across doses | 42 | 37 | 16
  Related Irritability, Across doses | 238 | 227 | 232
  Any Loss of appetite, Across doses | 155 | 145 | 153
  Grade 3 Loss of appetite, Across doses | 4 | 4 | 1
  Related Loss of appetite, Across doses | 152 | 144 | 148

39. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs) - Primary Vaccination.
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" is defined an incidence of an unsolicited AE regardless of intensity or relationship to study vaccination.
Time Frame: Within the 31-day (Days 0-30) post-primary vaccination
Population: The Primary Total Vaccinated cohort included all vaccinated subjects who received at least one primary dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 260 | 260 | 260
Participants | 181 | 177 | 185

40. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: Throughout the entire study period (up to Month 21)
Population: The Primary Total Vaccinated cohort included all vaccinated subjects who received at least one primary dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 260 | 260 | 260
Participants | 35 | 26 | 35

41. Secondary Outcome: Number of Subjects With Solicited Local Symptoms -Booster Vaccination
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any occurrence of the specified symptom regardless of intensity. Grade 3 pain was defined as cried when limb was moved/spontaneously painful. Grade 3 redness/swelling was defined as redness/swelling > 30 millimeters from injection site.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following booster dose
Population: The Booster Total Vaccinated cohort included all subjects vaccinated with the booster dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 257 | 258 | 258
Participants
  Any Pain | 174 | 161 | 145
  Grade 3 Pain | 21 | 21 | 7
  Any Redness | 175 | 144 | 180
  Grade 3 Redness | 22 | 10 | 10
  Any Swelling | 185 | 146 | 160
  Grade 3 Swelling | 27 | 15 | 11

42. Secondary Outcome: Number of Subjects With Solicited General Symptoms - Booster Vaccination.
Description: as for outcome 38
Time Frame: During the 4-day (Days 0-3) post-vaccination period following booster dose
Population: The Booster Total Vaccinated cohort included all subjects vaccinated with the booster dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 256 | 258 | 258
Participants
  Any Drowsiness | 131 | 118 | 128
  Grade 3 Drowsiness | 6 | 5 | 3
  Related Drowsiness | 126 | 110 | 121
  Any Temperature | 100 | 100 | 103
  Grade 3 Temperature | 1 | 2 | 1
  Related Temperature | 95 | 89 | 93
  Any Irritability | 167 | 161 | 166
  Grade 3 Irritability | 11 | 8 | 1
  Related Irritability | 161 | 147 | 159
  Any Loss of appetite | 93 | 83 | 111
  Grade 3 Loss of appetite | 5 | 0 | 2
  Related Loss of appetite | 89 | 72 | 101

43. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs) - Booster Vaccination.
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" was defined an incidence of an unsolicited AE regardless of intensity or relationship to study vaccination.
Time Frame: Within the 31-day (Days 0-30) after booster vaccination
Population: The Booster Total Vaccinated cohort included all subjects vaccinated with the booster dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
Number analyzed (Participants) | 257 | 259 | 258
Participants | 106 | 105 | 105

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Days 0-3) post-primary and post-booster vaccination; Unsolicited AEs: during the 31-day (Days 0-30) post-primary and post-booster vaccination; SAEs: during the entire study period (up to Month 21).
Arm/Group | Synflorix + Infanrix Hexa Group | Synflorix + Pediacel Group | Prevenar + Pediacel Group
All-Cause Mortality (participants affected / at risk) | 0/260 | 0/260 | 0/260
Serious Adverse Events (participants affected / at risk) | 35/260 | 26/260 | 35/260
Other Adverse Events (participants affected / at risk) | 260/260 | 260/260 | 260/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synflorix + Infanrix Hexa Group (N=260) | Synflorix + Pediacel Group (N=260) | Prevenar + Pediacel Group (N=260)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Velo-cardio-facial syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Adhesion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (3) | 0 (0)
Bronchiolitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 8 (8) | 4 (4) | 5 (5)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Pneumonia primary atypical (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 5 (5) | 2 (2) | 5 (5)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 2 (2)
Greenstick fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Feeding disorder neonatal (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 4 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synflorix + Infanrix Hexa Group (N=260) | Synflorix + Pediacel Group (N=260) | Prevenar + Pediacel Group (N=260)
Decreased appetite (Metabolism and nutrition disorders) | 182 (326) | 174 (309) | 191 (342)
Diarrhoea (Gastrointestinal disorders) | 22 (25) | 21 (24) | 15 (17)
Eczema (Skin and subcutaneous tissue disorders) | 25 (25) | 16 (17) | 18 (19)
Enteritis (Gastrointestinal disorders) | 17 (17) | 8 (9) | 12 (12)
Erythema (Skin and subcutaneous tissue disorders) | 231 (546) | 210 (528) | 222 (542)
Gastroenteritis (Infections and infestations) | 23 (24) | 17 (17) | 17 (17)
Injection site haematoma (General disorders) | 12 (15) | 16 (16) | 7 (8)
Irritability (Psychiatric disorders) | 252 (676) | 242 (659) | 247 (649)
Otitis media (Infections and infestations) | 22 (22) | 14 (14) | 10 (11)
Pain (General disorders) | 227 (573) | 219 (527) | 208 (464)
Pyrexia (General disorders) | 195 (364) | 179 (297) | 164 (275)
Somnolence (Nervous system disorders) | 240 (598) | 237 (544) | 225 (553)
Swelling (General disorders) | 232 (610) | 220 (559) | 211 (516)
Upper respiratory tract infection (Infections and infestations) | 117 (153) | 125 (160) | 133 (170)
Viral infection (Infections and infestations) | 10 (12) | 24 (24) | 10 (10)
Vomiting (Gastrointestinal disorders) | 13 (14) | 16 (20) | 10 (10)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 10 (11) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.